CLINICAL TRIAL: NCT05345093
Title: Open, Non-comparative, Multicentre, Interventional Clinical Investigation to Evaluate the Performance and Safety of the Medical Device Ialuxid® Gel (Hydrogen Peroxide and Hyaluronic Acid) in the Treatment of Acne Vulgaris and Folliculitis.
Brief Title: Evaluation of Safety and Performance of Ialuxid Gel in Treatment of Acne Vulgaris, and Folliculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BMG Pharma (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPBMG/0122/MD
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Acne Vulgaris; Folliculitis
MeSH Terms: conditions — Acne Vulgaris; Folliculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ialuxid Gel (Experimental): twenty-two patients affected by acne vulgaris; twenty-two patients affected by folliculitis.
  Interventions: Device: Ialuxid gel

INTERVENTIONS:
Device: Ialuxid gel — Ialuxid® Gel is intended for topical external use. It is formulated with the appearance of white to pale yellow coloured consistent gel.
  Ialuxid® Gel will be used for 8 weeks, 2-3 times a day.

SUMMARY:
The Research Question of the present study is the following: in a population of men and women affected by acne vulgaris, and folliculitis, will Ialuxid® Gel (hydrogen peroxide, hyaluronic acid and glycine) improve the course of the disease, resulting in a decrease of the total number of lesions, results observed after 4 and 8 weeks after the beginning of the treatment?

DETAILED DESCRIPTION:
Ialuxid® Gel is a non-antibiotic treatment in gel indicated for use in a variety of skin conditions, and also in case of infection. Its principal ingredient is Ialuvance™ Complex, a proprietary association of hydrogen peroxide, hyaluronic acid, and glycine.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 18 and ≤ 45 years.
2. Patients diagnosed with acne vulgaris, and folliculitis.

   a. Only for patients with acne vulgaris: mild to moderate Global Acne Grading Scale score (≤ 30).
3. Patients willing to provide signed informed consent to clinical investigation participation.
4. Patients who agree to discontinue all dermatological treatment and procedures during the study.
5. Patients able to communicate adequately with the Investigator and to comply with the requirements for the study.

Exclusion Criteria:

1. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study.

   *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
2. Patients with history of allergy or hypersensitivity to Hyaluronic Acid or to any other ingredients of Ialuxid® Gel or hypersensitivity skin reaction to Ialuxid® Gel based on skin test results.
3. History of anaphylaxis or severe complicated allergy symptoms.
4. Patients with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma.
5. Patients who have used oral drugs for acne vulgaris, and folliculitis in the previous month.
6. Patients who have used topical therapies for acne vulgaris, and folliculitis in the previous month.
7. Use of concomitant treatments or procedures aimed to improve skin condition over the last six months before the enrolment, such as chemical peeling, dermabrasion, laser resurfacing.
8. Patients suffering from infectious diseases that would compromise participation, including herpes simplex virus infection, active hepatitis, or human immunodeficiency virus.
9. Patients at risk in term of precautions, warnings and contra-indications referred in the package insert of Ialuxid® Gel.
10. Patients with any facial aesthetic surgery (such as facial contouring surgery: rhinoplasty, chin, or cheek enhancement (through facial implant) or facial rejuvenation surgery: facelift, eyelid lift, neck lift or facial implants etc.) in the preceding 3 months before the enrolment.
11. Patients who received filler injections of any typology in the face in the preceding 3 months.
12. Patients who received botulinum toxin A injections in the face in the preceding 6 months.
13. Need to have direct or indirect contact with quaternary ammonium salts during the study.
14. Patients unlikely to cooperate.
15. Patients with any other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalization during the study.
16. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change in total number of lesions | 8 weeks
  To evaluate the overall performance of the medical device Ialuxid Gel in the treatment of acne vulgaris, and folliculitis in terms of change in the total number of lesions, according to lesions count performed by Investigator (sum of lesions present on the body area mainly interested by each disease, to be specified in CRF).
Adverse event incidence | 8 weeks
  To evaluate the safety of the device trough Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Serious Adverse event incidence | 8 weeks
  To evaluate the safety of the device trough Serious Adverse Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Adverse Device event incidence | 8 weeks
  To evaluate the safety of the device trough Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Serious Adverse Device event incidence | 8 weeks
  To evaluate the safety of the device trough Serious Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Anticipated Serious Adverse Device event incidence | 8 weeks
  To evaluate the safety of the device trough Anticipated Serious Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation.
Unexpected Serious Adverse Device event incidence | 8 weeks
  To evaluate the safety of the device trough Unexpected Serious Adverse Device Event incidence assessed by Investigators at all visits and reported according to the current legislation.

SECONDARY OUTCOMES:
Change in total number of lesions | 4 weeks
  To evaluate the overall performance of the medical device Ialuxid® Gel in the treatment of acne vulgaris, and folliculitis in terms of change in the total number of lesions, according to lesions count performed by Investigator
Global Acne Grading System (GAGS) | 8 weeks
  To assess acne vulgaris severity by means of the Global Acne Grading System (GAGS) score, assessed by Investigator. Only for patients affected by acne vulgaris.
  The grading system score evaluates the acne severity from a minimum score of 0 (no acne) to >39 (very severe acne).
Total Severity Score (TSS) | 8 weeks
  To assess the total number of patients having a decrease in the global severity of the disease by means of the Total Severity Score (TSS), assessed by Investigator.
  The scale evaluates of symptoms of each diseases (for folliculitis - pustule and inflammatory nodules; for acne vulgaris - comedones, papules, pustules, nodules, cysts, abscesses) from 0 (absent) to 3 (severe).
Treatment satisfaction questionnaire | 8 weeks
  To assess the patient satisfaction by means of the treatment satisfaction questionnaire, assessed by patient, providing their degree of satisfaction with the treatment on a four-point scale (very satisfied, satisfied, moderately satisfied, or not satisfied)
Investigator Global Assessment of Performance (IGAP) | 8 weeks
  To evaluate the global performance of Ialuxid® Gel by means of the Investigator Global Assessment of Performance (IGAP), assessed by Investigator, through photos taken at each visit. The scale evaluates the change on a 4 point scale from 1 meaning very good performance to 4 meaning poor performance)
Investigator Global Assessment of Performance (IGAS) | 8 weeks
  To evaluate the global safety of Ialuxid® Gel by means of the Investigator Assessment of Performance (IGAS) assessed by the Investigator, providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.
Patient Global Assessment of Performance (PGAS) | 8 weeks
  To evaluate the global safety of Ialuxid® Gel by means of the Patient Assessment of Performance (PGAS) assessed by the patient, providing the safety on a four point scale from 4 meaning poor safety to 1 meaning very good safety.
Dermatology Life Quality Index (DLQI) | 8 weeks
  To assess the quality of life by means of the Dermatology Life Quality Index (DLQI) score, assessed by patients, providing the impact the disease had on the subjects life in various scenarios from not at all to very much

CONTACTS AND LOCATIONS:
Overall Officials: Petronela Mitrica, Principal Investigator — Salvosan-Ciobanca
Locations (1):
- SC Salvosan Ciobanca SRL, Zalău, Sălaj County, Romania

REFERENCES:
- [Background] Alsulaimani H, Kokandi A, Khawandanh S, Hamad R. Severity of Acne Vulgaris: Comparison of Two Assessment Methods. Clin Cosmet Investig Dermatol. 2020 Sep 28;13:711-716. doi: 10.2147/CCID.S266320. eCollection 2020. PMID 33061511
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008 Nov;159(5):997-1035. doi: 10.1111/j.1365-2133.2008.08832.x. Epub 2008 Sep 15. PMID 18795920
- [Background] Gravitz L. Skin. Nature. 2018 Nov;563(7732):S83. doi: 10.1038/d41586-018-07428-4. No abstract available. PMID 30464282
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? J Invest Dermatol. 2005 Oct;125(4):659-64. doi: 10.1111/j.0022-202X.2005.23621.x. PMID 16185263
- [Background] Inoue K, Takei K, Denda M. Functional glycine receptor in cultured human keratinocytes. Exp Dermatol. 2015 Apr;24(4):307-9. doi: 10.1111/exd.12651. PMID 25644897
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Kapoor P, Kumar S. Hydrogen peroxide in dermatology. Indian J Dermatol Venereol Leprol. 2023 Jan-Mar;89(2):310-312. doi: 10.25259/IJDVL_292_2021. No abstract available. PMID 34623047
- [Background] Keen MA. Hyaluronic Acid in Dermatology. Skinmed. 2017 Dec 1;15(6):441-448. eCollection 2017. PMID 29282181
- [Background] Khavkin J, Ellis DA. Aging skin: histology, physiology, and pathology. Facial Plast Surg Clin North Am. 2011 May;19(2):229-34. doi: 10.1016/j.fsc.2011.04.003. PMID 21763983
- [Background] Kim J, Ko Y, Park YK, Kim NI, Ha WK, Cho Y. Dietary effect of lactoferrin-enriched fermented milk on skin surface lipid and clinical improvement of acne vulgaris. Nutrition. 2010 Sep;26(9):902-9. doi: 10.1016/j.nut.2010.05.011. PMID 20692602
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Majtan J, Bucekova M, Jesenak M. Natural Products and Skin Diseases. Molecules. 2021 Jul 25;26(15):4489. doi: 10.3390/molecules26154489. PMID 34361642
- [Background] Nardi NM, Schaefer TJ Impetigo [Updated 2021 Aug 11]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2022 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK430974/
- [Background] NCBI Bookshelf. A service of the National Library of Medicine, National Institutes of Health. Clinical Review Report: Ozenoxacin 1% Cream (Ozanex): (Ferrer Internacional, S.A.): Indication: The topicaltreatment of impetigo in patients aged two months and older [Internet]. Ottawa (ON): Canadian Agency forDrugs and Technologies in Health; 2018 Oct
- [Background] Pereira H, Sousa DA, Cunha A, Andrade R, Espregueira-Mendes J, Oliveira JM, Reis RL. Hyaluronic Acid. Adv Exp Med Biol. 2018;1059:137-153. doi: 10.1007/978-3-319-76735-2_6. PMID 29736572
- [Background] Reddy J, Rao V, Madhavulu B et al A randomized open label parallel group study comparing the safety, effectiveness and adherence between 2% fusidic acid cream versus 1% retapamulin ointment in children with impetigo International Journal of Basic & Clinical Pharmacology February 2019
- [Background] Salwowska NM, Bebenek KA, Zadlo DA, Wcislo-Dziadecka DL. Physiochemical properties and application of hyaluronic acid: a systematic review. J Cosmet Dermatol. 2016 Dec;15(4):520-526. doi: 10.1111/jocd.12237. Epub 2016 Jun 21. PMID 27324942
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jul 15;59(2):e10-52. doi: 10.1093/cid/ciu444. PMID 24973422
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] Sutaria AH, Masood S, Saleh HM, Schlessinger J. Acne Vulgaris. 2023 Aug 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459173/ PMID 29083670
- [Background] Veraldi S, Micali G, Berardesca E, Dall'Oglio F, Sinagra JL, Guanziroli E. Results of a Multicenter, Randomized, Controlled Trial of a Hydrogen Peroxide-based Kit versus a Benzoyl Peroxide-based Kit in Mild-to-moderate Acne. J Clin Aesthet Dermatol. 2016 Oct;9(10):50-54. Epub 2016 Oct 1. PMID 27847549
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- [Background] Winters RD, Mitchell M Folliculitis [Updated 2021 Aug 11]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2022 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK547754/
- [Derived] Stefancu ME, Barattini DF, Botnaru I, Vizman C, Stucchi L, Barattini L. Performance and Safety of the Medical Device Ialuxid Gel in the Treatment of Mild-Moderate Acne Vulgaris: An Open-Label, Noncomparative Multicentre Interventional Clinical Trial. J Cosmet Dermatol. 2025 Mar;24(3):e70084. doi: 10.1111/jocd.70084. PMID 40029154